CLINICAL TRIAL: NCT06427564
Title: Vital Signs Data Collection Using "Comestai" Application
Brief Title: Vital Signs Collection Via "Comestai" App
Status: Recruiting | Type: Observational
Sponsor: Buzzi Children's Hospital (Other)
Responsible Party: Principal Investigator, Valeria Calcaterra, Clinical Professor, Buzzi Children's Hospital
Other Study IDs: CET 98-2024
Record Dates: First submitted 2024-05-15; First posted 2024-05-24 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Vital Signs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to verify and validate the parameters collected from mobile devices via the app named "Comestai" and from reference devices. The assessments considered to define comorbidities are included.. Specifically, collection of vital parameters (Blood Pressure, Heart Rate, Respiratory Rate, Oxygen Saturation) through the "Comestai" Application via mobile phones (using photoplethysmographic method) and reference devices such as Withings-Blood Pressure Monitor Connect® (for Blood Pressure), Polar Verity Sense® (for Heart Rate), Masimo-finger sensor® (for Oxygen Saturation, Respiratory Rate), comparing and confirming them. Consent will be sought for the viewing and collection of blood test results that are normally included in evaluations for subjects with overweight and/or obesity and/or diabetes.

Estimated time required for each measurement recording: 10-15 minutes per subject

Total number of subjects: 3000

DETAILED DESCRIPTION:
Early detection of variations in vital parameters allows for the identification of changes in patients' health status and the provision of recommendations for therapeutic adjustments. The application named "Comestai" is a non-invasive and easy-to-use tool that enables the measurement of vital parameters. The app allows users to simultaneously measure vital parameters such as Heart Rate (HR), Respiratory Rate (RR), Oxygen Saturation (SpO2), and Blood Pressure (BP) using the photoplethysmographic method with the front camera of a mobile device.

The use of simultaneous vital parameter measurement systems like apps can enhance self-monitoring of health status and improve patient care. In this study, vital parameters will be measured using the "Comestai" application and compared and validated with measurements from standard clinical practice devices.

Consent will be sought for the viewing and collection of biochemical evaluation results typically required for individuals with overweight and/or obesity and/or diabetes.

"Comestai" Application: This wellness app allows for non-invasive measurement of vital parameters, enabling users to detect SpO2, HR, RR, and BP by looking at the front camera of a mobile device ("By Face"). The measurement method used is Remote Photoplethysmography (rPPG).

This is a prospective, open-label, study to collect vital parameters using the Comestai application by looking at the front camera of a mobile device ("By Face"). The measurement method of the app is Remote Photoplethysmography (rPPG).

The study plans to enroll up to 3000 subjects

Each subject will be assigned a specific identification number (Subject ID). During the evaluation, the following data will be recorded in the Electronic Case Report Form (eCRF):

Medical history of the subject Current or past therapies Demographic data (date of birth, sex) Smoking habits Physical characteristics (height in meters, weight in kilograms, Body Mass Index in kg/m^2, and phototype)

During the 'By Face' measurement of vital parameters with the app, subjects will be asked to sit in a comfortable place, looking at the phone screen (about 25 cm away) with their face fully uncovered (no masks, hats, or any facial accessories). During data collection, the subject should remain still and breathe steadily. The subject will be required to look directly at the camera throughout the data collection process. The 'By Face' data collection mode can be performed on both iOS and Android in parallel, with both devices positioned in front of the subject. HR and blood pressure will also be measured immediately before and after the app measurement.

Data Collection Equipment

For vital signs data collection using the "Comestai" application, the study staff will use the following mobile phones for rPPG "By Face" measurements:

* Face: Apple internet(i)Phone 13 Pro (10 bit) & Samsung Galaxy S21 Ultra
* Two additional phones will be used as remote:
* One Android phone - Recorder Remote to start the measurement from far.
* One Apple iPhone -Masimo-finger sensor App to collect the data from the Masimo finger sensor.
* Other necessary equipment includes phone stands (two per room of measurement). In addition to the equipment for vital signs data collection using the "Comestai" application, reference devices will measure the subject's vital signs as a point of comparison.

rPPG "By Face" vital signs data collection includes videoing the subjects' faces with a mobile device (iOS and Android) front camara for approximately 1.5 minutes.

Vital signs data using the reference devices (i.e., SpO2, RR, BP, PR) will be collected continuously for approximately 1.5 minutes, and simultaneously to the data collected using the "Comestai" application (i.e., "By Face").

Several data collection events (1.5 minutes each) may be performed per subject using the "Comestai" application and reference devices.

BP will be collected using the reference devices prior to data collection using the Comestai application and immediately after completion of data collection using the Comestai application.

During "By Face" data collection, the subjects will be requested to sit in a comfortable place, looking at a screen (distance of ~25cm) with a fully exposed face (not to wear a mask, hat, or any kind of accessory on the face). During data collection, the subject breathing should be stable with minimum movements. The subject will be requested to stare directly towards the camara during the whole data collection process.

"By Face" mode of data collection can be taken for both iOS and Android in parallel when both devices are positioned in front of the subject.

During the "By Face" data collection, SpO2 levels will be monitored continuously using the standard reference device.

Consent will be sought for viewing and collecting the results of pre-scheduled blood tests. Participation is optional, and subjects who do not consent can still proceed with the parameter measurements. In case of acceptance, the following results will be considered:

Complete Blood Count (Hemoglobin, White Blood Cell Count, Neutrophils, Lymphocytes, and Platelets), Hemoglobin Glycosylated (HbA1C), Lipid Profile (Total Cholesterol, Cholesterol-LDL, Cholesterol-HDL, and Triglycerides), Glucose, Alanine transaminase (ALT), Creatinine.

Estimated participation time per subject: approximately 10-15 minutes.

No medical decisions will be based on data obtained through the "Comestai" application, reference devices, or blood sample results.

All data will be recorded in the study's eCRF.

The analysis plan involves verifying and validating the parameters collected from mobile devices via the app and from reference devices, as well as results of pre-scheduled blood tests and patient demographic data. For all parameters, the accuracy of the app measurement compared to the reference device and standard tests will be assessed.

Confidence intervals will be calculated using the bootstrap method. The correlation between measurements using the app and those using reference devices and standard tests will be evaluated using the Pearson correlation coefficient. The agreement between the two measurements (app and reference devices/and standard tests) will be represented using Bland-Altman plots.

ELIGIBILITY:
Inclusion Criteria:

Prior to enrollment in this study, subjects must meet all the following inclusion criteria:

1. Subject must have the ability to understand and provide written informed consent.
2. Male or Female subject ≥16 and ≤65 of age.
3. Subject must be willing and able to comply with study procedures.

Exclusion Criteria:

Subjects will be excluded from the study if any of the following conditions are present:

1. Subject with compromised circulation, injury, or physical malformation of fingers, hands, ears or forehead/skull or other sensor Region of Interest (ROI) which would limit the ability to test ROI needed for the study.
2. Subject has a tattoo in the optical path which would limit the ability to test ROI needed for the study.
3. Subjects with severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, respiration monitor electrodes or other medical sensors used for measuring vital signs.
4. Subject with a medical condition which in the opinion of the investigator, does not allow performing the study assessments.
5. Subject unfit to participate in the study to the judgment of the investigator.

In addition to the Inclusion/Exclusion criteria, the 70% of target population should include adult subjects with at least one of the following:

* Pre-diabetes or diabetes HbA1C 5.7-13%
* >30% of subjects with HbA1C 5.7-6.4%
* >30% of subjects with HbA1C >6.4%
* Hypertension with systolic measurements above 130 mmHg
* >40% of subjects with systolic BP >130 mmHg
* >20% of subjects with systolic BP >160 mmHg
* Total cholesterol: >40% of subjects with >200 mg/dl and/or LDL above 130 mg/dl
* Atrial fibrillation 1%
* Smokers ~ 20-30% of all subjects in the study

Note: the same subject can have more than one of the above medical conditions. It is preferred that subjects will be treatment- naive for the medical condition they suffer from or are not under treatment at the time of participation (e.g. a subject who suffers from hypertension has not started his treatment to lower his blood pressure).

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Potential adolescent and adult subjects (male and female ≥16 and ≤65 of age), of any race, physiques and skin pigmentation with awide range of health conditions who provided their consent by signing the informed consent form will be screened into the study and provided with a subject specific identification number used throughout the study (i.e. Subject ID).
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Data Collection Storage and Processing-Pulse rate | 15 minutes for data collection
  Collect, verify and validate Pulse rate (beats per minute) in data using the Comestai application and reference devices.
  Pulse rate data obtained using the Comestai application and reference data will be stored on Comestai's secured cloud without any subject identifiable information and will only be recognized using the subject identification number provided during screening. The raw data of subjects' vital signs will be locked, encrypted, and can be read only by Study center team.
  The measurement method utilized by the app is Remote Photoplethysmography (rPPG).
  No medical decisions will be made based on the data obtained using the Comestai application, the reference devices, and the pre-scheduled blood sample results.
Data Collection Storage and Processing-Oxygen saturation | 15 minutes for data collection
  Collect, verify and validate Oxygen saturation (percentage) in data using the Comestai application and reference devices.
  Oxygen saturation data obtained using the Comestai application and reference data will be stored on Comestai's secured cloud without any subject identifiable information and will only be recognized using the subject identification number provided during screening. The raw data of subjects' vital signs will be locked, encrypted, and can be read only by Study center team.
  The measurement method utilized by the app is Remote Photoplethysmography (rPPG).
  No medical decisions will be made based on the data obtained using the Comestai application, the reference devices, and the pre-scheduled blood sample results.
Data Collection Storage and Processing-Respiratory rate | 15 minutes for data collection
  Collect, verify and validate Respiratory rate (breaths per minute) in data using the Comestai application and reference devices.
  Respiratory rate data obtained using the Comestai application and reference data will be stored on Comestai's secured cloud without any subject identifiable information and will only be recognized using the subject identification number provided during screening. The raw data of subjects' vital signs will be locked, encrypted, and can be read only by Study center team.
  The measurement method utilized by the app is Remote Photoplethysmography (rPPG).
  No medical decisions will be made based on the data obtained using the Comestai application, the reference devices, and the pre-scheduled blood sample results.
Data Collection Storage and Processing-Blood pressure | 15 minutes for data collection
  Collect, verify and validate Blood pressure (mmHg) in data using the Comestai application and reference devices.
  Blood pressure data obtained using the Comestai application and reference data will be stored on Comestai's secured cloud without any subject identifiable information and will only be recognized using the subject identification number provided during screening. The raw data of subjects' vital signs will be locked, encrypted, and can be read only by Study center team.
  The measurement method utilized by the app is Remote Photoplethysmography (rPPG).
  No medical decisions will be made based on the data obtained using the Comestai application, the reference devices, and the pre-scheduled blood sample results.

SECONDARY OUTCOMES:
Data Collection Storage and Processing-Hemoglobin | 15 minutes for data collection
  Collect, verify and validate Hemoglobin level (g/dl) in data using the Comestai application and results of pre-scheduled blood tests
  Hemoglobin level data obtained using the Comestai application and results of pre-scheduled blood tests will be stored on Comestai's secured cloud without any subject identifiable information and will only be recognized using the subject identification number provided during screening. The raw data of subjects' vital signs will be locked, encrypted, and can be read only by Study center team.
  The measurement method utilized by the app is Remote Photoplethysmography (rPPG).
  No medical decisions will be made based on the data obtained using the Comestai application, the reference devices, and the pre-scheduled blood sample results.
Data Collection Storage and Processing-Hemoglobin glycosylated | 15 minutes for data collection
  Collect, verify and validate Hemoglobin glycosylated level (mmol/mol) in data using the Comestai application and results of pre-scheduled blood tests
  Hemoglobin glycosylated level data obtained using the Comestai application and and results of pre-scheduled blood tests will be stored on Comestai's secured cloud without any subject identifiable information and will only be recognized using the subject identification number provided during screening. The raw data of subjects' vital signs will be locked, encrypted, and can be read only by Study center team.
  The measurement method utilized by the app is Remote Photoplethysmography (rPPG).
  No medical decisions will be made based on the data obtained using the Comestai application, the reference devices, and the pre-scheduled blood sample results.

CONTACTS AND LOCATIONS:
Overall Officials: Gianvincenzo Zuccotti, MD, Prof, Principal Investigator — Buzzi Children's Hospital
Locations (1):
- ASST-Fatebenefratelli Sacco-Buzzi Children's Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zuccotti G, Agnelli PO, Labati L, Cordaro E, Braghieri D, Balconi S, Xodo M, Losurdo F, Berra CCF, Pedretti RFE, Fiorina P, De Pasquale SM, Calcaterra V. Vital Sign and Biochemical Data Collection Using Non-contact Photoplethysmography and the Comestai Mobile Health App: Protocol for an Observational Study. JMIR Res Protoc. 2025 Apr 28;14:e65229. doi: 10.2196/65229. PMID 40293779